CLINICAL TRIAL: NCT01278628
Title: SUMCO Metabolic Syndrome Project
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Fukuoka University (Other)
Responsible Party: Principal Investigator, Yuichiro Nishida, Lecturer, Fukuoka University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 19200049sagasumco
Record Dates: First submitted 2011-01-18; First posted 2011-01-19 (Estimated); Last update posted 2016-08-10 (Estimated); Status verified 2016-08

CONDITIONS: Metabolic Syndrome
MeSH Terms: conditions — Metabolic Syndrome | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Lifestyle modification (Experimental)
  Interventions: Other: exercise training

INTERVENTIONS:
Other: exercise training — exercise class once a year

SUMMARY:
Physical activity is considered important in prevention and treatment of obesity and metabolic syndrome. Genotype of genes involved in metabolism is also known to be associated with the development of metabolic syndrome. However, scarce evidence exists regarding the influence of physical activity intensity and genotype on metabolic syndrome in people with obesity. The investigators examine physical activity using an uniaxial accelerometer, as well as aerobic fitness using an electric bicycle ergometer, several genotypes of genes related to glucose and lipid metabolisms in middle-aged men with obesity and/or abdominal obesity who were employees in silicon wafer manufacture and participated in a health checkup.

ELIGIBILITY:
Inclusion Criteria:

* healthy people and individuals with obesity and metabolic syndrome

Exclusion Criteria:

-

Ages: 40 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2009-08; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Components of metabolic syndrome | every year

CONTACTS AND LOCATIONS:
Locations (1):
- SUMCO corporation, Imari, Saga-ken, Japan